CLINICAL TRIAL: NCT03828682
Title: A 12-Month, Open Label Study of Extended Release Tacrolimus (Envarsus XR®, LCPT) With Mycophenolate, Rabbit Antithymocyte Globulin (rATG) and Early Steroid Withdrawal in de Novo Kidney Transplant Recipients
Brief Title: Veloxis de Novo Kidney Transplant ECSWD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simon Tremblay, PharmD, PhD (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Simon Tremblay, PharmD, PhD, Research Assistant Professor of Surgery, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-7742
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Kidney Transplantation; Immunosuppression
Keywords: tacrolimus; extended release; kidney transplantation; steroid withdrawal; once daily
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Methylprednisolone; Prednisone; thymoglobulin

STUDY DESIGN:
Intervention Model Description: A prospective cohort of de novo kidney transplant recipients will be assigned to treatment group and compared to historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective Arm (Experimental): De novo kidney transplant recipients receiving:
  rabbit antithymocyte globulin induction (1.5mg/kg, dosage range 4-6mg/kg total dose over 5-10 days) 5-day steroid withdrawal (methylprednisolone 500mg IV on day 1 (day of transplant), 250mg IV on day 2, 125mg IV on day 3, prednisone 80mg PO on day 4, 60mg PO on day 5 and then no more steroids Once-daily tacrolimus XR 0.8mg/kg/day started when or when serum creatinine is <4mg/dL or by 48 hours of transplant to target 24-hr trough levels of 8-12ng/mL up to day 30 followed by 24-hour trough targets of 5-10ng/mL Mycophenolate mofetil (1000 mg PO BID) or mycophenolic acid (720mg PO BID) twice daily started prior to surgery
  Interventions: Drug: Tacrolimus Extended Release Oral Tablet [Envarsus]; Drug: Mycophenolate Mofetil; Drug: Mycophenolic Acid Oral Product; Drug: Methylprednisolone; Drug: Prednisone; Drug: Rabbit Anti-Human T-Lymphocyte Globulin Injectable Solution [Thymoglobulin]
- Comparator arm (Active Comparator): Historical control arm consisting of the following
  De novo kidney transplant recipients receiving:
  rabbit antithymocyte globulin induction (1.5mg/kg, dosage range 4-6mg/kg total dose over 5-10 days) 5-day steroid withdrawal (methylprednisolone 500mg IV on day 1 (day of transplant), 250mg IV on day 2, 125mg IV on day 3, prednisone 80mg PO on day 4, 60mg PO on day 5 and then no more steroids Twice-daily tacrolimus 0.1mg/kg/day started when or when serum creatinine is <4mg/dL or by 48 hours of transplant to target 12-hr trough levels of 8-12ng/mL up to day 30 followed by 12-hour trough targets of 5-10ng/mL Mycophenolate mofetil (1000 mg PO BID) or mycophenolic acid (720mg PO BID) twice daily started prior to surgery
  Interventions: Drug: Mycophenolate Mofetil; Drug: Mycophenolic Acid Oral Product; Drug: Tacrolimus; Drug: Methylprednisolone; Drug: Prednisone; Drug: Rabbit Anti-Human T-Lymphocyte Globulin Injectable Solution [Thymoglobulin]

INTERVENTIONS:
Drug: Tacrolimus Extended Release Oral Tablet [Envarsus] — Tacrolimus Extended Release Oral Tablet [Envarsus]
  Other Names: Envarsus XR
  Arms: Prospective Arm
Drug: Mycophenolate Mofetil — Mycophenolate mofetil capsules or tablets
  Other Names: Cellcept; MMF
Drug: Mycophenolic Acid Oral Product — mycophenolic acid tablets
  Other Names: Myfortic; MPA
Drug: Tacrolimus — Twice daily tacrolimus
  Other Names: Prograf; FK506
  Arms: Comparator arm
Drug: Methylprednisolone — Methylprednisolone taper
Drug: Prednisone — Prednisone taper
  Other Names: Deltasone
Drug: Rabbit Anti-Human T-Lymphocyte Globulin Injectable Solution [Thymoglobulin] — Rabbit Anti-Human T-Lymphocyte Globulin
  Other Names: Thymoglobulin; rATG

SUMMARY:
This study is designed to evaluate the safety and efficacy of LCPT in combination with rATG, mycophenolate and early corticosteroid withdrawal (CSWD) in de novo kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 18 years of age.
2. Patient who is receiving a renal transplant from a living or heart-beating deceased donor.
3. Female patients of child bearing potential must have a negative urine or serum pregnancy test within the past 48 hours prior to study inclusion.
4. The patient has given written informed consent to participate in the study

Exclusion Criteria:

1. Patient has previously received an organ transplant other than a kidney.
2. Patient is receiving an HLA identical living donor transplant.
3. Patient who is a recipient of a multiple organ transplant.
4. Patient has a most recent cytotoxic PRA of >25% or calculated PRA >50% where multiple moderate level HLA antibodies exist and in the opinion of the PI represents substantial HLA sensitization.
5. Patient with a positive T or B cell crossmatch that is primarily due to HLA antibodies.
6. Patient with a donor specific antibody (DSA) as deemed by the PI to be associated with significant risk of rejection.
7. Patient has received an ABO incompatible donor kidney.
8. The deceased donor and/or deceased donor kidney meet any of the following extended criteria for organ donation (ECD):

   1. Donor age ≥ 60 years OR
   2. Donor age 50-59 years and 1 of the following:

   i. Cerebrovascular accident (CVA) + hypertension + SCr > 1.5 mg/dL OR ii. CVA + hypertension OR iii. CVA + SCr > 1.5 mg/dL OR iv. Hypertension + SCr > 1.5 mg/dL OR c. CIT ≥ 24 hours, donor age > 10 years OR d. Donation after cardiac death (DCD)
9. Recipients will be receiving a dual or en bloc kidney transplant.
10. Donor anticipated cold ischemia is >30hours.
11. Recipient that is seropositive for hepatitis C virus (HCV) with detectable Hepatitis C viral load are excluded. HCV seropositive patients with a negative HCV viral load testing may be included.
12. Recipients with a positive hepatitis B viral load or positive hepatitis B surface antigen testing within 1 year of consent.
13. Hepatitis B surface antibody negative recipients receiving a kidney from a donor seropositive for hepatitis B core antibody or hepatitis B nucleic acid.
14. Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV).
15. Recipient who is seronegative for Epstein Barr Virus (EBV)
16. Patient has uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives.
17. Patients with thrombocytopenia (PLT <75,000/mm3), and/or leukopenia (WBC < 2,000/mm3), or anemia (hemoglobin < 6 g/dL) prior to study inclusion.
18. Patient is taking or has been taking an investigational drug in the 30 days prior to transplant.
19. Patient who has undergone desensitization therapy within 6 months prior to transplant.
20. Patient has a known hypersensitivity to tacrolimus, mycophenolate mofetil/mycophenolic acid, rabbit anti-thymocyte globulin, or glucocorticoids.
21. Patient is receiving chronic steroid therapy at the time of transplant.
22. Patients with a history of cancer (other than non-melanoma skin cell cancers cured by local resection) within the last 5 years, unless they have an expected disease free survival of >95%.
23. Patient is pregnant, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by positive human Chorionic Gonadotropin (hCG) laboratory test.
24. Women of childbearing potential must use reliable contraception simultaneously, unless they are status post bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.
25. Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.
26. Inability to cooperate or communicate with the investigator.
27. Renal allograft has been reperfused for more than 48 hours at the time of enrollment
28. Patient unable to receive intact LCPT formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with the combination oral outcome of Biopsy-proven acute rejection, patient death and graft loss | 12 months
  Biopsy-proven acute rejection, patient death and graft loss

CONTACTS AND LOCATIONS:
Overall Officials: Simon Tremblay, PharmD, PhD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No